CLINICAL TRIAL: NCT04001699
Title: Interprofessional Preoperative Geriatric Assessment for Older Arthroplasty Patients With Multimorbidity - a Randomized Clinical Trial
Brief Title: Interprofessional Preoperative Geriatric Assessment for Older Arthroplasty Patients With Multimorbidity
Acronym: IPPGA-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Eastern Finland (Other)
Collaborators: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Eija Lönnroos, professor, University of Eastern Finland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HERIT
Record Dates: First submitted 2019-06-25; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Multimorbidity; Knee Arthrosis; Hip Arthrosis
Keywords: preoperative; geriatric assessment; interprofessional team
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Preoperative assessment conducted by an interprofessional team
  Interventions: Other: Preoperative geriatric assessment
- Usual care (Active Comparator): Usual care
  Interventions: Other: Preoperative geriatric assessment

INTERVENTIONS:
Other: Preoperative geriatric assessment — In addition to the usual care, patients randomized to the intervention group receive preoperative assessment conducted by an interprofessional team including geriatrician, registered nurse, physiotherapist and pharmacist. Based on the assessment, a preoperative optimization plan is constructed focusing on the treatment of the patient's chronic conditions, nutritional status, medication and physical activity.

SUMMARY:
The objective of this randomized control trial is to investigate effects and cost effectiveness of interprofessional preoperative assessment among older knee or hip arthroplasty patients. The main hypothesis is that preoperative assessment and optimization have a positive impact on the patents' quality of life and expenditure of social and health care services.

DETAILED DESCRIPTION:
Knee and hip arthrosis are common conditions among older adults. Progression of arthrosis often leads to worsening of symptoms and decreased mobility, daily functioning and quality of life. Total joint arthroplasty improves pain in end-stage arthrosis but accustomed postoperative care and rehabilitation alone may not guarantee optimal regain of functioning for frail and vulnerable older arthroplasty patients. Preoperative optimization of older patients with multimorbidity and functional limitations may improve benefits of the arthroplasty even at lower costs. Patients randomized into intervention arm of the present study receive preoperative assessment with treatment and prehabilitation plan. The focuses of the intervention are patient's chronic conditions, nutritional status, medication and physical activity. The intervention is delivered by multiprofessional team (geriatrician, registered nurse, physiotherapist and pharmacist).

Older adults undergoing surgery are a rapidly growing but vulnerable patient group. Knowledge on effects of preoperative evaluation and optimization is sparse, especially on the effects of multi-domain interventions.

ELIGIBILITY:
Inclusion Criteria:

* Place of residence: Kuopio or Vesanto municipality
* Age ≥ 65 years
* Clinical decision for knee or hip arthroplasty, elective operation with more than one month waiting time, primary arthroplasty of the index joint.
* Multimorbidity: the patient has at least two chronic diseases with potential to affect functioning, diseases are defined according to the Function Comorbidity Index (FCI)

Additional inclusion criteria, at least two of the following:

* 5 or more medicines taken regularly (polypharmacy)
* continuous walking distance less than 500 m
* needs help in dressing and/or washing oneself
* needs help when visiting or taking care of businesses outside home
* body mass index ≤ 23 or ≥ 34

Exclusion Criteria:

- does not meet the above inclusion criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-08-19 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life (15-D) | Preoperative measurement at baseline, postoperative measurements 3 and 9 months after the arthroplasty.
  Change in quality of life is measured using the 15-dimensions health-related quality of life questionnaire (15-D) in three time points
Costs of social and health care services | Changes in costs of care are evaluated for a period starting from one year before and ending two years after the baseline examinations.
  Data on the use and costs of social and health care services are obtained from the national and local care registers. The costs of the intervention are evaluated by measuring working time of the inter-professional team members (used per every study patient).

CONTACTS AND LOCATIONS:
Overall Officials: Eija Lönnroos, Principal Investigator — University of Eastern Finland, Institute of Public Health and Clinical Nutrition
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No